CLINICAL TRIAL: NCT01827046
Title: Minimally Invasive Surgery Plus Rt-PA for ICH Evacuation Phase III
Acronym: MISTIE-III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Genentech, Inc. (Industry); Emissary International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00080619; U01NS080824 (NIH); ICH02 (Other: Other)
Record Dates: First submitted 2013-04-01; First posted 2013-04-09 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: intracerebral hemorrhage; ICH; brain hemorrhage; minimally invasive surgery; rt-PA
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MIS plus rt-PA management (Experimental): Subjects randomized to the Minimally Invasive Surgery (MIS) plus rt-PA management arm will undergo minimally invasive surgery followed by up to 9 doses of 1.0 mg of rt-PA (Activase/Alteplase/CathFlo) for intracerebral hemorrhage clot resolution.
  Interventions: Drug: rt-PA
- Medical management (No Intervention): Subjects randomized to medical management will receive the standard medical therapies for the treatment of intracerebral hemorrhage, which includes ICU care only and no planned surgical intervention.

INTERVENTIONS:
Drug: rt-PA — Up to 9 doses of 1.0 mg of rt-PA will be administered through the catheter that was placed directly into the intracerebral hemorrhage using minimally invasive surgery.
  Other Names: Activase; Alteplase; CathFlo
  Arms: MIS plus rt-PA management

SUMMARY:
A phase III, randomized, case-controlled, open-label, 500-subject clinical trial of minimally invasive surgery plus rt-PA in the treatment of intracerebral hemorrhage (ICH).

DETAILED DESCRIPTION:
Primary Objectives:

Efficacy: Demonstrate that minimally invasive surgery (MIS) plus recombinant tissue plasminogen activator (rt-PA) for three days improves functional outcome by a 12% increase in the modified Rankin Scale (mRS) score 0-3 compared to medically treated subjects assessed at 365 days.

Secondary Objective:

Demonstrate that the end of treatment volume and percent of ICH reduction from MIS+rt-PA is related to improved functional outcome, as compared to medically treated subjects.

Safety:

Demonstrate that early use of MIS+rt-PA for three days is safe for the treatment of ICH relative to rates of mortality, rebleeding, and infection in the medically treated subject at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous supratentorial ICH ≥ 30 mL diagnosed using radiographic imaging (computerized tomography (CT), computerized tomography angiography (CTA), etc.), with a Glasgow Coma Scale (GCS) ≤ 14 or a NIHSS ≥ 6.
* Stability CT scan done at least 6 hours after diagnostic CT showing clot stability (growth < 5 mL as measured by ABC/2 method).
* Symptoms less than 24 hours prior to diagnostic CT (dCT) scan (an unknown time of onset is exclusionary).
* Ability to randomize between 12 and 72 hours after dCT.
* Systolic Blood Pressure (SBP) < 180 mmHg sustained for six hours recorded closest to the time of randomization.
* Historical Rankin score of 0 or 1.
* Age ≥ 18 and older.

Exclusion Criteria:

* Infratentorial hemorrhage.
* Intraventricular hemorrhage (IVH) requiring treatment for IVH-related (casting) mass effect or shift due to trapped ventricle. External ventricular drain (EVD) to treat intracranial pressure (ICP) is allowed.
* Thalamic bleeds with apparent midbrain extension with third nerve palsy or dilated and non-reactive pupils. Other (supranuclear) gaze abnormalities are not exclusions. Note: Patients with a posterior fossa ICH or cerebellar hematomas are ineligible.
* Irreversible impaired brain stem function (bilateral fixed, dilated pupils and extensor motor posturing), GCS ≤ 4.
* Ruptured aneurysm, arteriovenous malformation (AVM), vascular anomaly, Moyamoya disease, hemorrhagic conversion of an ischemic infarct, recurrence of a recent (< 1 year) hemorrhage diagnosed with radiographic imaging.
* Patients with unstable mass or evolving intracranial compartment syndrome.
* Platelet count < 100,000; international normalized ratio (INR) > 1.4.
* Any irreversible coagulopathy or known clotting disorder.
* Inability to sustain INR ≤ 1.4 using short- and long-active procoagulants (such as but not limited to NovoSeven, Fresh Frozen Plasma (FFP), and/or vitamin K).
* Subjects requiring long-term anti-coagulation are excluded. Reversal of anti-coagulation is permitted for medically stable patients who can realistically tolerate the short term risk of reversal. Patient must not require Coumadin (anticoagulation) during the first 30 days, and normalized coagulation parameters must be demonstrated, monitored closely and maintained during the period of brain instrumentation.
* Use of Dabigatran, Apixaban, and/or Rivaroxaban (or a similar medication from the similar medication class) prior to symptom onset.
* Internal bleeding, involving retroperitoneal sites, or the gastrointestinal, genitourinary, or respiratory tracts.
* Superficial or surface bleeding, observed mainly at vascular puncture and access sites (e.g., venous cutdowns, arterial punctures, etc.) or site of recent surgical intervention.
* Positive urine or serum pregnancy test in pre-menopausal female subjects without a documented history of surgical sterilization.
* Allergy/sensitivity to rt-PA.
* Prior enrollment in the study.
* Participation in a concurrent interventional medical investigation or clinical trial. Patients in observational, natural history, and/or epidemiological studies not involving an intervention are eligible.
* Not expected to survive to the day 365 visit due to co-morbidities and/or are do not resuscitate (DNR)/ do not intubate (DNI) status prior to randomization.
* Any concurrent serious illness that would interfere with the safety assessments including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease.
* Patients with a mechanical heart valve. Presence of bio-prosthetic valve(s) is permitted.
* Known risk for embolization, including history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* In the investigator's opinion, the patient is unstable and would benefit from a specific intervention rather than supportive care plus or minus MIS+rt-PA removal of the ICH.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2013-12-30 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F. Hanley, MD, Study Chair — Johns Hopkins University; Mario Zuccarello, MD, Principal Investigator — University of Cincinnati; Issam Awad, MD, Principal Investigator — University of Chicago
Locations (84):
- United States (56):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mercy San Juan Medical Center, Carmichael, California
  - Scripps Health, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Stanford University, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Northshore University Health System, Evanston, Evanston, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Heath System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - University of Buffalo, Buffalo, New York
  - North Shore Long Island Jewish Health System, Manhasset, New York
  - Mount Sinai Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - State University of New York, Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Providence Brain and Spine Institute, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern at Dallas, Dallas, Texas
  - University of Texas, Houston, Houston, Texas
  - University of Texas at San Antonio, San Antonio, Texas
  - Intermountain Neurosciences Institute, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Fairfax INOVA Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Adelaide Hospital, North Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - McMaster University, Hamilton, Ontario
  - Montreal Neurological Institute, McGill University, Montreal, Quebec
- China (3):
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Bayi Brain Hospital, Beijing Military General Hospital, Beijing
  - Southwest Hospital, Third Military Medical University, Chongqing
- Germany (4):
  - University of Bonn, Bonn
  - University of Heidelberg, Heidelberg
  - University of Mainz, Mainz
  - University of Munich, Munich
- Hungary (3):
  - University of Pecs, Pécs, Baranya
  - University of Debrecen, Debrecen
  - University of Szeged, Szeged
- Israel (2):
  - The Chaim Sheba Medical Center at Tel Hashomer, Tel Litwinsky, Ramat-Gan
  - Rabin Medical Center, Petah Tikva
- Spain (6):
  - Hospital Universitario Cruces, Barakaldo, Biscay
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Bellvitge, Barcelona
  - Hospital Universitario Mutua de Terrassa, Barcelona
  - Hospital Universitario Rio Hortega, Valladolid
- United Kingdom (4):
  - Salford Royal NHS Foundation Trust, Salford, Manchester
  - South Glasgow University Hospital, Glasgow
  - Newcastle Royal Victoria Infirmary, Newcastle upon Tyne
  - University of Southampton Hospital, Southampton

REFERENCES:
- [Derived] Cooper DC, Abramson E, Ziai WC, Flaherty ML, Shah VA, Avadhani R, Ostapkovich N, Carhuapoma L, Awad I, Zuccarello M, Hanley D, Sansing LH. Intracerebral haemorrhage laterality and associations with mood and pain: a MISTIE III substudy. Stroke Vasc Neurol. 2025 Dec 23;10(6):734-742. doi: 10.1136/svn-2024-003755. PMID 40250866
- [Derived] Sun P, Badihian S, Avadhani R, Walborn N, Yarava A, Alimoradi D, Awad I, Hanley D, Murthy S, Ziai W. Does stereotactic thrombolysis with alteplase for intracerebral haemorrhage alter intraventricular haematoma volume? A secondary analysis of the MISTIE-III trial. J Neurol Neurosurg Psychiatry. 2024 Sep 17;95(10):892-898. doi: 10.1136/jnnp-2023-333032. PMID 38670789
- [Derived] Bako AT, Potter T, Pan AP, Tannous J, Britz G, Ziai WC, Awad I, Hanley D, Vahidy FS. Minimally Invasive Surgery With Thrombolysis for Intracerebral Hemorrhage Evacuation: Bayesian Reanalysis of a Randomized Controlled Trial. Neurology. 2023 Oct 17;101(16):e1614-e1622. doi: 10.1212/WNL.0000000000207735. Epub 2023 Sep 8. PMID 37684058
- [Derived] Magid-Bernstein JR, Li Y, Cho SM, Piran PJ, Roh DJ, Gupta A, Shoamanesh A, Merkler A, Zhang C, Avadhani R, Montano N, Iadecola C, Falcone GJ, Sheth KN, Qureshi AI, Rosand J, Goldstein J, Awad I, Hanley DF, Kamel H, Ziai WC, Murthy SB. Cerebral Microbleeds and Acute Hematoma Characteristics in the ATACH-2 and MISTIE III Trials. Neurology. 2022 Mar 8;98(10):e1013-e1020. doi: 10.1212/WNL.0000000000013247. Epub 2021 Dec 22. PMID 34937780
- [Derived] Hanley DF, Thompson RE, Rosenblum M, Yenokyan G, Lane K, McBee N, Mayo SW, Bistran-Hall AJ, Gandhi D, Mould WA, Ullman N, Ali H, Carhuapoma JR, Kase CS, Lees KR, Dawson J, Wilson A, Betz JF, Sugar EA, Hao Y, Avadhani R, Caron JL, Harrigan MR, Carlson AP, Bulters D, LeDoux D, Huang J, Cobb C, Gupta G, Kitagawa R, Chicoine MR, Patel H, Dodd R, Camarata PJ, Wolfe S, Stadnik A, Money PL, Mitchell P, Sarabia R, Harnof S, Barzo P, Unterberg A, Teitelbaum JS, Wang W, Anderson CS, Mendelow AD, Gregson B, Janis S, Vespa P, Ziai W, Zuccarello M, Awad IA; MISTIE III Investigators. Efficacy and safety of minimally invasive surgery with thrombolysis in intracerebral haemorrhage evacuation (MISTIE III): a randomised, controlled, open-label, blinded endpoint phase 3 trial. Lancet. 2019 Mar 9;393(10175):1021-1032. doi: 10.1016/S0140-6736(19)30195-3. Epub 2019 Feb 7. PMID 30739747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and randomization occurred at 78 hospitals in USA, Canada, Europe, Australia, and Asia
Groups:
- MIS Plus Rt-PA Management: Subjects randomized to the Minimally Invasive Surgery (MIS) plus recombinant tissue plasminogen activator (rt-PA) management arm will undergo minimally invasive surgery followed by up to 9 doses of 1.0 mg of rt-PA (Activase/Alteplase/CathFlo) for intracerebral hemorrhage clot resolution.
  rt-PA: Up to 9 doses of 1.0 mg of rt-PA will be administered through the catheter that was placed directly into the intracerebral hemorrhage using minimally invasive surgery.
Period: Overall Study
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Started | 250 | 249
Completed | 249 | 240
Not Completed | 1 | 9
Not completed — Lost to Follow-up | 1 | 5
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- MIS Plus Rt-PA Management: Subjects randomized to the MIS plus rt-PA management arm will undergo minimally invasive surgery followed by up to 9 doses of 1.0 mg of rt-PA (Activase/Alteplase/CathFlo) for intracerebral hemorrhage clot resolution.
  rt-PA: Up to 9 doses of 1.0 mg of rt-PA will be administered through the catheter that was placed directly into the intracerebral hemorrhage using minimally invasive surgery.
- Total: Total of all reporting groups
Arm/Group | MIS Plus Rt-PA Management | Medical Management | Total
Number analyzed (Participants) | 250 | 249 | 499
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [52 to 70] | 62 [53 to 71] | 62 [52 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 103 | 194
  Male | 159 | 146 | 305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 34 | 68
  Not Hispanic or Latino | 216 | 215 | 431
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 12 | 18 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 46 | 41 | 87
  White | 190 | 184 | 374
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Australia | 2 | 2 | 4
  Canada | 3 | 4 | 7
  China | 5 | 5 | 10
  Europe | 41 | 44 | 85
  United States | 199 | 194 | 393
Tobacco use [Count of Participants; unit: Participants] | 50 | 39 | 89
Cocaine use [Count of Participants; unit: Participants] | 11 | 9 | 20
On anticoagulants [Count of Participants; unit: Participants] | 24 | 10 | 34
Hormone replacement therapy [Count of Participants; unit: Participants] | 1 | 3 | 4
Hyperlipidaemia medication compliant [Count of Participants; unit: Participants] | 96 | 93 | 189
Antiplatelet therapy [Count of Participants; unit: Participants] | 67 | 77 | 144
Diabetes [Count of Participants; unit: Participants] | 72 | 67 | 139
Hypertension [Count of Participants; unit: Participants] | 241 | 240 | 481
Other cardiovascular disease [Count of Participants; unit: Participants] | 38 | 34 | 72
GCS score at randomization [Count of Participants; unit: Participants] — Glasgow Coma Scale (GCS) scores range from 15 (fully conscious) to 3 (Deep coma)
  Participants
    3-8 | 64 | 63 | 127
    9-12 | 111 | 108 | 219
    13-15 | 75 | 78 | 153
NIHSS score at randomization [Median (Inter-Quartile Range); unit: Units on a scale] — NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The maximum possible score is 42, with the minimum score being a 0. Stroke severity is scored in the following way:0=No stroke symptoms,1-4=Minor stroke, 5-15=Moderate stroke,16-20=Moderate to severe stroke, 21-42=Severe stroke
  Units on a scale | 19 [15 to 23] | 19 [15 to 23] | 19 [15 to 23]
Diagnostic CT at presentation - IntraCerebral Hemorrhage (ICH) volume (mL) [Median (Inter-Quartile Range); unit: mL] | 42.7 [30.4 to 54.5] | 41.5 [30.9 to 55.3] | 41.8 [30.8 to 54.5]
Diagnostic CT at presentation - IntraVentricular Hemorrhage (IVH) volume (mL) [Median (Inter-Quartile Range); unit: mL] | 0 [0 to 1.7] | 0 [0 to 1.9] | 0 [0 to 1.9]
Stability CT(last CT before randomization) IntraCerebral Hemorrhage (ICH) volume (mL) [Median (Inter-Quartile Range); unit: mL] | 45.8 [35.4 to 59.6] | 45.3 [35.4 to 57.2] | 45.6 [35.6 to 58.7]
Stability CT(last CT before randomization) IntraVentricular Hemorrhage (IVH) volume (mL) [Median (Inter-Quartile Range); unit: mL] | 0.3 [0 to 3.1] | 0.4 [0 to 3.2] | 0.4 [0 to 3.2]
Ventilated at randomization [Count of Participants; unit: Participants] | 107 | 102 | 209
Blood pressure at presentation [Median (Inter-Quartile Range); unit: mm Hg]
  Systolic BP (mm Hg) | 177 [155 to 208] | 176 [158 to 200] | 177 [156 to 204]
  Diastolic BP (mm Hg) | 99 [85 to 113] | 98 [84 to 114] | 98 [84 to 113]
Blood pressure at randomization [Median (Inter-Quartile Range); unit: mm Hg]
  Systolic BP (mm Hg) | 138 [130 to 148] | 138 [131 to 148] | 138 [131 to 148]
  Diastolic BP (mm Hg) | 70 [63 to 78] | 69 [60 to 77] | 69 [62 to 77]
Time from stroke to diagnostic CT (h) [Median (Inter-Quartile Range); unit: Hours] | 2.2 [1.1 to 6.0] | 1.9 [1.2 to 4.8] | 2.0 [1.2 to 5.1]
Time from stroke to stability CT (h) [Median (Inter-Quartile Range); unit: Hours] | 36.4 [23.4 to 52.6] | 36.3 [23.6 to 48.6] | 36.3 [23.5 to 50.2]
Clot location [Count of Participants; unit: Participants]
  Deep | 163 | 144 | 307
  Lobar | 87 | 105 | 192
mRS score before stroke [Count of Participants; unit: Participants] — Score 0 = No symptoms. Score 1 = Having symptoms but no significant disability, and is able to carry out all usual activities.
  Participants
    0 | 230 | 233 | 463
    1 | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Dichotomized, Adjudicated Modified Rankin Scale Score 0-3 vs. 4-6 at 365 Days Post Ictus (Adjusted)
Description: Dichotomized, adjudicated, cross-sectional modified Rankin Scale (mRS) score 0-3 vs. 4-6 at 365 days post-ictus, adjusting for baseline (pre-randomization) variables used in covariate adaptive randomization as well as the clinically established severity variables IVH size and ICH location (lobar or deep). Ictus refers to symptom onset.
  The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death. Dichotomized scores are: 0-3=No symptoms to moderate disability requiring some assistance; 4-6=Moderately severe disability requiring complete assistance to death.
Time Frame: Day 365
Population: Includes participants with mRS scores available at day 365. Number and proportions reported refer to number of participants and proportions with Modified Rankin Score 0-3
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 249 | 240
Participants
  mRS 0-3 | 110 | 100
  mRS 4-6 | 139 | 140
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.73, Chi-squared; Risk Difference (RD) = 2, 95% CI 2-sided [-6.8 to 10.7]
Statistical Analysis 2: Comparison: MIS Plus Rt-PA Management vs Medical Management; Adjusted for age, GCS, stability ICH volume, stability IVH volume, ICH deep location; Test type: Superiority; p = 0.33, Multivariate logit model; Risk Difference (RD) = 4, 95% CI 2-sided [-4 to 12]

2. Secondary Outcome: Dichotomized Extended Glasgow Outcome Scale (eGOS) Score UGR-US vs. LS-Death at 365 Days Post Ictus (Adjusted)
Description: Dichotomized, cross-sectional extended Glasgow Outcome Scale (eGOS) score upper good recovery (UGR) through upper severe disability (US) vs. lower severe disability (LS) through death at 365 days post ictus, adjusting for baseline (pre-randomization) variables used in covariate adaptive randomization as well as the clinically established severity variables IVH size and ICH location (lobar or deep).
  The eGOS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored as: 1=Death, 2=Vegetative state, 3=Lower severe disability, 4=Upper severe disability, 5=Lower moderate disability, 6=Upper moderate disability, 7=Lower good recovery, 8=Upper good recovery. Dichotomous variable coding is as follows: 1=codes 4-8, 0=codes 1-3.
Time Frame: Day 365
Population: Those with non-missing mRS scores at 365 days post ictus
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 244 | 234
Participants
  eGOS UGR-US (4-8) | 94 | 84
  eGOS LS-Death (1-3) | 150 | 150
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.55, Chi-squared; Risk Difference (RD) = 0.03, 95% CI 2-sided [-0.06 to 0.11]
Statistical Analysis 2: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.27, Multivariate logit model; Adjusted for age, GCS, stability ICH volume, stability IVH volume and ICH deep location; Risk Difference (RD) = 1.26, 95% CI 2-sided [0.82 to 1.97]

3. Secondary Outcome: All Cause Mortality Longitudinally From Ictus to 365 Days (Adjusted)
Description: By group comparison of mortality from ictus to 365 days adjusted for baseline severity.
Time Frame: Day 365
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Participants | 48 | 62
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.08, Log Rank
Statistical Analysis 2: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.037, Adjusted Cox proportional Hazard; Adjusted for age, GCS, Stability ICH volume, Stability IVH volume, ICH deep location, diabetes, cardiovascular disease and race; Cox Proportional Hazard = 0.67, 95% CI 2-sided [0.45 to 0.98]

4. Secondary Outcome: Clot Removal (Amount of Residual Blood)
Description: Relationship between clot removal as an Area Under the Curve (AUC) clot-assessment that estimates the time-averaged clot volume from ictus to end of treatment (EOT i.e. 24 hours after last dose) as AUC clot exposure and functional outcome (proportion 0-3 Modified Rankin Scale (mRS)).
Time Frame: 24 hours after last dose
Population: Includes patients who survived through the dosing period
Measure: Mean (Standard Deviation); unit: 10mL x days
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 246 | 239
10mL x days
  mRS 0-3 | 2.69 (1.11) | 4.11 (1.35)
  mRS 4-6 | 3.32 (1.33) | 5.26 (1.82)
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p < 0.001, Logit model; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.62 to 0.80]
Statistical Analysis 2: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p < 0.001, Multivariate logit model; Adjusted for age, GCS, stability IVH volume, and ICH deep location; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.59 to 0.78]

5. Secondary Outcome: Patient Disposition: Home Days Over 365 Days Time From Ictus.
Description: By group comparison of cumulative days at home during the 365 days post ictus.
Time Frame: During 365 days of follow-up
Population: Includes only patients with cumulative home days at any time during the 365 days of follow-up.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 166 | 157
Days | 306 [237 to 329] | 300 [232 to 328]
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Patient Disposition: Patient Location at 365 Days Post Ictus (i.e., Good vs. Bad Location) (Adjusted)
Description: Patient disposition: By group comparison of residential location at day 365 post ictus adjusted for baseline severity.
  Good locations refers to home and rehabilitation; and bad locations refers to acute care, long-term care and death.
Time Frame: Day 365
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Participants
  Good Location | 163 | 151
  Bad location | 87 | 98
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.34, Chi-squared; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.04 to 0.11]

7. Secondary Outcome: Dichotomized, Adjudicated, Cross-sectional Modified Rankin Scale (mRS) Score 0-3 vs. 4-6 180 Days Post Ictus (Adjusted)
Description: Dichotomized, adjudicated, cross-sectional modified Rankin Scale (mRS) score 0-3 vs. 4-6 at 180 days post-ictus, adjusting for baseline (pre-randomization) variables used in covariate adaptive randomization as well as the clinically established severity variables IVH size and ICH location (lobar or deep).
  The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death. Dichotomized scores are: 0-3=No symptoms to moderate disability requiring some assistance; 4-6=Moderately severe disability requiring complete assistance to death
Time Frame: Day 180
Population: Includes patients who were not lost to followup at day 180
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 243
Participants
  mRS 0-3 | 99 | 93
  mRS 4-6 | 151 | 150
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.76, Chi-squared; Risk Difference (RD) = -0.01, 95% CI 2-sided [-0.10 to 0.07]
Statistical Analysis 2: Comparison: MIS Plus Rt-PA Management; Test type: Superiority; p = 0.31, Multivariate logit model; Adjusted for age, GCS, Stability ICH volume, Stability IVH volume, ICH deep location; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.81 to 1.94]

8. Secondary Outcome: Dichotomized Extended Glasgow Outcome Scale (eGOS) Score UGR-US vs. LS-Death at 180 Days Post Ictus (Adjusted)
Description: Dichotomized, cross-sectional extended Glasgow Outcome Scale (eGOS) score upper good recovery (UGR) through upper severe disability (US) vs. lower severe disability (LS) through death at 180 days post ictus, adjusting for baseline (pre-randomization) variables used in covariate adaptive randomization as well as the clinically established severity variables IVH size and ICH location (lobar or deep).
  The eGOS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored as: 1=Death, 2=Vegetative state, 3=Lower severe disability, 4=Upper severe disability, 5=Lower moderate disability, 6=Upper moderate disability, 7=Lower good recovery, 8=Upper good recovery. Dichotomous variable coding is as follows: 1=codes 4-8, 0=codes 1-3.
Time Frame: Day 180
Population: Patients were included if they were not lost to followup at day 180
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 243
Participants
  eGOS UGR-US (4-8) | 81 | 76
  eGOS LS-Death (1-3) | 169 | 167
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management; Test type: Superiority; p = 0.79, Chi-squared; Risk Difference (RD) = 0.01, 95% CI 2-sided [-0.07 to 0.09]
Statistical Analysis 2: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.35, Multivariate logit model; Adjusted for age, GCS, Stability ICH volume, Stability IVH volume, ICH deep location; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.79 to 1.97]

9. Secondary Outcome: Type and Intensity of ICU Management: ICU Days
Description: By group comparison of cumulative number of days in the Intensive Care Unit (ICU) in a hospital
Time Frame: Up to 365 days
Population: Includes patients with cumulative ICU days during the 365 days of follow-up
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 240 | 238
Days | 10 [7 to 17] | 10 [5 to 16]
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.46, Median test

10. Secondary Outcome: Type and Intensity of ICU Management: Hospital Days
Description: By group comparison of total number of days in the hospital
Time Frame: Up to 365 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Days | 17 [13 to 27] | 17 [10 to 25]
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.75, Median test

11. Secondary Outcome: EQ-VAS
Description: By group comparison of EQ-VAS at day 365 post ictus. The EuroQol Visual Analogue Scale (EQ-VAS) is a self-reported measure of health status. It is a marked scale where subjects draw a line to indicate their health, with end points of 0 (the worst health you can imagine) and 100 (the best health you can imagine).
Time Frame: Day 365
Population: Includes patients who survived or were not lost to followup through 365 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 183 | 164
score on a scale | 70 [50 to 80] | 70 [50 to 80]
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: EuroQol 5 Dimensional Scale (EQ-5D)
Description: By group comparison of EQ-5D at day 365 post ictus. The EuroQol 5 Dimensional Scale (Eq-5D) is a self-reported measure of health status. It is arranged to assess domains related to mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each domain, codes were 1=no problems, 2=some problems, 3=extreme problems, and 9=unknown. Having a problem in at least 1 domain was coded as 1 (originally represented by 2 or 3) and no problems as 0 (originally represented by 1) .
Time Frame: Day 365
Population: Patients were included if they survived or were not lost to followup through 365 days
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 192 | 170
Participants
  Any problem | 176 | 155
  No problem | 16 | 15
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.87, Chi-squared

13. Other Pre Specified Outcome: Mortality and Safety Events: First-week (Operative) Mortality
Description: Mortality and Safety events: By group comparison of mortality within the first 7 days post randomization.
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Participants | 2 | 10
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.02, Chi-squared

14. Other Pre Specified Outcome: Mortality and Safety Events: All Cause Mortality
Description: By group comparison of mortality from all causes within the first 30 days post randomization.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Participants | 23 | 37
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.05, Chi-squared

15. Other Pre Specified Outcome: Mortality and Safety Events: Adjudicated Symptomatic Brain Bleeding Within 72 Hours After Last Dose
Description: By group comparison of the percentage of subjects experiencing one or more adjudicated symptomatic brain bleeding events within the first 30 days post randomization.
Time Frame: 72 hours after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Participants | 6 | 3
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.32, Chi-squared

16. Other Pre Specified Outcome: Mortality and Safety Events: Adjudicated Bacterial Brain Infection
Description: By group comparison of the percentage of subjects experiencing one or more adjudicated brain bacterial infection events within the first 30 days post randomization.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Participants | 2 | 0
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.16, Chi-squared

17. Other Pre Specified Outcome: Mortality and Safety Events: Total Serious Adverse Events (SAE) at 30 Days
Description: By group comparison of the total number of adjudicated serious adverse events that occurred within the first 30 days post randomization.
Time Frame: Day 30
Measure: Number; unit: Number of events
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Number of events | 123 | 136
Statistical Analysis 1: Comparison: MIS Plus Rt-PA Management vs Medical Management; Test type: Superiority; p = 0.01, Chi-squared

18. Other Pre Specified Outcome: Mortality and Safety Events: Summary of AE and SAE by MedDRA Code and Grouped by Organ System Within the First 30 Days Post Ictus
Description: By group comparison of the total number of adjudicated adverse events (AE) and serious adverse events (SAE) across all coded organ systems that occurred within the first 30 days post ictus.
Time Frame: Day 30
Measure: Number; unit: Number of events
Arm/Group | MIS Plus Rt-PA Management | Medical Management
Number analyzed (Participants) | 250 | 249
Number of events
  Serious Adverse Events | 123 | 136
  Adverse Events | 477 | 378

ADVERSE EVENTS:
Time Frame: 30 days post-ictus
Arm/Group | MIS Plus Rt-PA Management | Medical Management
All-Cause Mortality (participants affected / at risk) | 48/250 | 62/249
Serious Adverse Events (participants affected / at risk) | 75/250 | 84/249
Other Adverse Events (participants affected / at risk) | 205/250 | 169/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIS Plus Rt-PA Management (N=250) | Medical Management (N=249)
Cardiac disorders (Cardiac disorders) | 3 (4) | 1 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (4) | 4 (6)
General disorders and administration site conditions (General disorders) | 13 (13) | 26 (27)
Non-neurological infections (Infections and infestations) | 2 (5) | 4 (8)
Injury, Poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasms(Benign, malignant or unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 17 (41) | 33 (62)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 1 (2)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (4)
Respiratory, thoracic and mediastinal disirders (Respiratory, thoracic and mediastinal disorders) | 26 (40) | 14 (25)
Vascular disorders (Vascular disorders) | 6 (11) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIS Plus Rt-PA Management (N=250) | Medical Management (N=249)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Cardiac disorders (Cardiac disorders) | 3 (15) | 5 (11)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (12) | 7 (17)
General disorders and administration site conditions (General disorders) | 17 (53) | 12 (42)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 2 (2)
Immune system disorders (Immune system disorders) | 0 (0) | 1 (1)
Infections, non-neurologic (Infections and infestations) | 9 (16) | 25 (41)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (4) | 2 (3)
Investigations (Investigations) | 1 (12) | 7 (20)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (17) | 6 (20)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Neoplasms: benign, malignant, Unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Nervous system disorders (Nervous system disorders) | 108 (216) | 47 (107)
Psychiatric disorders (Psychiatric disorders) | 6 (14) | 5 (13)
Renal and urinary disorders (Renal and urinary disorders) | 3 (5) | 2 (5)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 30 (67) | 33 (62)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Vascular disorders (Vascular disorders) | 14 (39) | 13 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT01827046/SAP_002.pdf
  • Study Protocol (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT01827046/Prot_003.pdf